CLINICAL TRIAL: NCT04484766
Title: Preeclampsia Associated Vascular Age- Long-term Follow-up and New Prevention Strategy
Brief Title: Preeclampsia Associated Vascular Aging
Acronym: PAVA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jena University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1498
Record Dates: First submitted 2020-04-15; First posted 2020-07-24 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient after pre-eclampsia: Patients with pre-eclampsia who were treated at the University Hospital of Jena between 1999-2009.
  Interventions: Other: Primary data collection
- Patients after PETN treatment: Patients of the PETN pilot study, with PETN and patients who received PETN as an individual therapy trial
  Interventions: Other: Primary data collection

INTERVENTIONS:
Other: Primary data collection — Primary data collection takes place via questionnaires outside the study centre.
  All other investigations take place at the study centre:
  * Physical examination: height, weight, BMI, blood pressure
  * Cardiac examination: cardiac output
  * Vascular measurements: Carotid intima media thickness, total peripheral resistance, blood pressure, flow-mediated vascular dilatation, critical flicker frequency, pulse wave velocity, augmentation index
  * Serum analysis: basic laboratory, multiplex analysis (human vascular inflammation, human angiogenesis and adhesion molecule panel)
  Other Names: Physical examination; Cardiac measurement; Vascular Measurement; Serum analysis

SUMMARY:
To evaluate cardiovascular health, especially endothelial health, of women after pre-eclampsia compared to women without pre-eclampsia, and to compare women who had taken PETN during pregnancy with women who had not attempted treatment

DETAILED DESCRIPTION:
The clinical observation that women with pre-eclampsia have a high risk of early onset cardiovascular disease with increased disease-associated mortality has led to the hypothesis that the endothelial status of these women is characterized by early onset of aging. We want to investigate the relationship between endothelial aging and pregnancy disorders such as pre-eclampsia, which are dominated by endothelial dysfunction. Do endothelial changes precede pregnancy and cause pre-eclampsia and later accelerated cardiovascular aging, or does pre-eclampsia trigger premature endothelial aging in affected individuals for the first time? The aim of this study is to investigate the cardiovascular health of women 10 to 20 years after pre-eclampsia and to compare it with that of women with uneventful pregnancies. In addition, the potential long-term endothelial protective effect of the NO-donor pentaerithrityltetranitrate (PETN) is investigated.

This in vivo study will be extended in vitro by the analysis of senescence induction in endothelial cells after pre-eclampsia associated stress. Additionally, the potential protective effect of PETN on stress-induced senescence will be evaluated.

The ultimate goal is to establish a prospective long-term study on the effect of PETN on vascular health in women with pre-eclampsia to assess whether treatment of endothelial dysfunction during pregnancy could reduce endothelial aging and thus premature cardiovascular morbidity and mortality in millions of women.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the PETN pilot study from 2002-2008
* controls: uneventful pregnancies from 2002-2008
* Patients with pre-eclampsia with PETN treatment 10-20 years ago
* Controls: patients with pre-eclampsia without PETN treatment 10-20 years ago
* Written Informed Consent
* Singleton pregnancy

Exclusion criteria:

* Patients who refuse to participate in the study
* Impossibility of the outpatient presentation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pre-eclampsia 10 to 20 years ago. The patients are matched with the next consenting patient who gave birth without pregnancy complications. Only singleton pregnancies born between the 24th and 42nd week of pregnancy are considered.
  Patients with and without PETN treatment are recruited from the patients who participated in the PETN pilot study from 2002 to 2008. In addition, patients are recruited who received PETN treatment as a personalised therapy trial. These are matched by patients without treatment. The matching includes the indication for treatment, the week of pregnancy at diagnosis and the percentiles of fetal growth
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
vascular health as combined outcome | 1 day 10-20 years after pregnancy
  Comparison of the vascular health of patients after pre-eclampsia with that of women with complication-free pregnancies 10-20 years after pregnancy by assessing physical parameters (height, weight, Blood pressure, bioelectric impedance analysis), measuring cardiac output, transthoracic echocardiography, carotid intima media thickness, total vascular resistance, flow mediated dilation, critical flicker frequency, puls-wave velocity and augmentation index
Potential long-term effect of PETN treatment using combined outcome of vascular health measurements in correlaation with treatment with PETN | 1 day 10-20 years after pregnancy
  Analysis of a possible long-term effect of PETN treatment during pregnancy based on a vascular health comparison of patients who received PETN in the PETN pilot study from 2002 to 2008, or who received it in a personalised therapy trial, with those who received placebo or no therapy
Endothelial cell senescence using senescence characterization of young and treated HUVEC cells | 1 day 10-20 years after pregnancy
  In vitro analysis of endothelial cell senescence established by hosting group after pre-eclampsia induced stress effect, as well as the possible protective effect of PETN on endothelial cell aging

CONTACTS AND LOCATIONS:
Overall Officials: Anna Multhaup, Dr. med., Principal Investigator — Klinik für Geburtsmedizin
Locations (1):
- Universitätsklinikum Jena, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No